CLINICAL TRIAL: NCT03134456
Title: Pembrolizumab for Metastatic Non-small Cell Lung Cancer (NSCLC) Patients Expressing PD-L1 Who Have Their Own Patient-derived Xenograft (PDX): Comparative Study of Clinical Response and In-vivo Antitumor Response Using Their Humanized CD34 PDX (Hu-CD34 PDX)
Brief Title: Pembrolizumab for Metastatic NSCLC Patients Expressing PD-L1 Who Have Their Own PDX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-004
Record Dates: First submitted 2017-04-06; First posted 2017-05-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm: pembrolizumab Injection (Experimental): Pembrolizumab according to the dosage and administration in Product Information of Keytruda in Korea (2mg/kg) until it is changed to 200mg flat dose.
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — Pembrolizumab according to the dosage and administration in Product Information of Keytruda in Korea (2mg/kg) until it is changed to 200mg flat dose.

SUMMARY:
This is a single center, open-label, single arm study in patients with metastatic non-small cell lung cancer (NSCLC) expressing PD-L1 after failure of platinum-based combination chemotherapy.

Patients will be treated with Pembrolizumab according to the dosage and administration in Product Information of Keytruda in Korea (2mg/kg) until it is changed to 200mg flat dose.

The patient should have their-own patient-derived xenograft (PDX) before enrollment of the study. The PDX will be used to set up their humanized CD34 PDX (Hu-CD34 PDX).

DETAILED DESCRIPTION:
Part A: Clinical trial (single arm study) in patients with metastatic non-small cell lung cancer (NSCLC) expressing PD-L1 after failure of platinum-based combination chemotherapy.

Part B: PDX experiment using Hu-CD34 PDX model in specific population selected from Part A (Clinical trial part) - responder and non-responder.

In-vivo experiment using Hu-CD34 PDX will be done for about seven subjects, and thirty-two (32) Hu-CD34 PDX mice will be established from single patient to see in-vivo response. This research using PDX (Part B) will be conducted sequentially on clinical trial part in selected-population based on clinical response of Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Have metastatic non-small cell lung cancer, which should be proven histologically.
3. Disease progression on or after platinum-based chemotherapy. Patients with sensitive EGFR mutations should have disease progression on at least one of EGFR TKIs (including but not limited to gefitinib, erlotinib, afatinib, osimertinib). Patients with ALK fusion should have disease progression on at least one of ALK TKI (including but not limited to crizotinib or ceritinib).

   a. Previously treated with 3 or more systemic regimens given for recurrent and/or metastatic disease are excluded (TKIs are not included in the number of regimens)
4. Have tumor which express PD-L1(TPS ≥ 1%) confirmed by immunohistochemistry.
5. Have their-own patient-derived xenograft established.
6. Over 18 years of age on day of signing informed consent.
7. Have measurable disease based on RECIST 1.1.
8. Have a performance status of 0 to 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.
12. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.7.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Hypersensitivity to pembrolizumab or any of its excipients.
4. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
7. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Evidence of interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B or Hepatitis C.
18. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Comparison of clinical response and in-vivo anti-tumor response using Hu-CD34 PDX | every 6 weeks, up to 96weeks
  response rate based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: sehoon lee, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No